CLINICAL TRIAL: NCT00334490
Title: A Phase II, Double Blind Randomized Controlled Trial to Determine the Safety and Efficacy of 12.5mg of Oral Sildenafil (Viagra) Compared to Placebo to Decrease Pulmonary Hypertension in Cardiac Patients After Cardiopulmonary Bypass
Brief Title: Does Oral Sildenafil (Viagra) Decrease Mean Pulmonary Artery Pressure After Cardiac Surgery?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 091532; REB 04-093 (Other: St Michael's Hospital, Toronto)
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Sildenafil; Viagra; Cardiac Surgery; Cardiopulmonary Bypass
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Oral Sildenafil 12.5 mg
  Interventions: Drug: Sildenafil
- 2 (Placebo Comparator): Placebo in 5 mls distilled water
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — 12.5 mg Sildenafil once with optional second dose
  Other Names: Viagra
  Arms: 1
Drug: Sildenafil — 12.5 mg orally once with optional second dose
  Other Names: Viagra
  Arms: 1
Drug: Placebo — Oral Placebo in 5 mls distilled water
  Other Names: Viagra
  Arms: 2

SUMMARY:
Post-operative pulmonary hypertension is a risk factor for right ventricular failure and an increasing cause of morbidity and mortality in patients undergoing high-risk cardiac surgery. Several treatments have been used to treat and reduce post operative pulmonary hypertension. Unfortunately none of these treatments are approved for use in this condition and only one (inhaled nitric oxide) is specific enough to pulmonary hypertension to not cause dangerous low blood pressure in the rest of the body. Sadly, inhaled nitric oxide is difficult and expensive to use, and can cause lung damage. Sildenafil citrate is quite specific to the lung vessels, is easy to administer and does not easily cause low blood pressure in other areas of the body. We hypothesize that oral sildenafil 12.5mg will decrease the baseline (pre-dose) mPAP by at least 20% compared with a placebo.

DETAILED DESCRIPTION:
Sildenafil citarte is a selective pulmonary vasodilator without profound effects on systemic hemodynamics making it an attractive option for treating post operative pulmonary hypertension in the cardiac surgical patients. It is inexpensive and feasible to administer. Intravenous as well as oral doses have been shown to reduce the mean pulmonary arterial pressure (mPAP) and pulmonary vascular resistance (PVR) in animal models as well as in clinical trials with adults with primary pulmonary hypertension and children after cardiac surgery . However, no data exists to support the safety and efficacy of Sildenafil citrate in the adult cardiac surgical population. The purpose of this study is to further investigate the potential role of Sildenafil citrate to treat post operative pulmonary hypertension in the cardiac population.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Scheduled for or has recently undergone a primary or re-do cardiac surgical procedure including coronary artery bypass graft surgery (CABG), heart valve replacement or repair, ascending aortic replacement or repair or any combinations of these procedures with CPB
* No documented allergy to sildenafil citrate
* No clinical or laboratory evidence on routine blood work of significant renal disease or failure. (requires dialysis or a creatinine >/= 200umol/L)
* No clinical or documented laboratory evidence on routine blood work of hepatic disease or failure. (ALT or AST 5x upper limit of normal (ULN) or jaundice)
* The patient if female and of child bearing age is not known to be pregnant.
* No documented history of severe chronic respiratory disease defined as an FEV/VC1< 50% predicted.
* Not currently enrolled as an active participant in another clinical trial of a medical therapy or device.
* No documented stroke or transient ischemic attack within 6 months of study participation
* No documented critical carotid artery stenosis (>70%)
* No retinitis pigmentosa.
* The patient has authorized his/her consent to participate in this trial pre-operatively OR consent to participation is granted on the patient's behalf by a substitute decision maker pre or post operatively.

POST-OPERATIVELY

* A pulmonary arterial catheter (swan-ganz catheter) is insitu.
* The patient has a mPAP measurement of >/= 25mmHg for at least 1 hour.
* The patient has a mean arterial pressure (MAP) of >/= 65mmHg.
* The patient has a heart rate of greater than 40 and less than 130 beats/minute.
* The patient is intubated and mechanically ventilated as per standard ventilation protocol at St. Michael's Hospital.
* The patient has not received intravenous nitroglycerin or nitroprusside within 1 hour before treatment with study medication.

Exclusion Criteria:

POST-OPERATIVELY

* The patient requires nitroglycerin based medications continuously (topical/oral/intravenous)
* The patient has an arterial pH of < 7.30 or ≥ 7.47
* The patient has clinical and or documented laboratory evidence from routine blood work of renal dysfunction or failure. (Doubling of pre-operative creatinine or requiring dialysis is indicative of renal dysfunction.)
* The patient has clinical and or documented laboratory evidence from routine blood work of significant hepatic disease or failure. (ALT or AST 5 times ULN or obvious jaundice will be indicative of liver dysfunction)
* The patient's current medical condition in the opinion of the investigator and/or the patient's attending ICU physician makes him/her inappropriate for participation in this study.
* The patient is currently a participant in a clinical trial of an investigational therapy including a drug or medical device.
* The patient has clinical indications of sepsis defined as 2 of the following five criteria: i) leukocytosis (or) leukopenia: wbc >12 x 109/L (or) <4x109/L (>10% bands also, ii) fever (or) hypothermia (temp >38.5C or <36C), iii) tachycardia, hr > 90 beats/minute, iv) tachypnea, respiratory rate (RR) >18 breaths/minute, v) hypotension, SBP <90 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-03; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of 12.5mg oral sildenafil to decrease the mPAP in patients presenting with a mPAP >/= 25mmHg after cardiopulmonary bypass. | Begining 2 hours postoperatively through 75 minutes post dosing

SECONDARY OUTCOMES:
To determine the efficacy of a second dose of oral sildenafil 12.5mg to decrease the mPAP in those patients who do not respond with a 20% decrease in mPAP after the initial administration of study medication. | From post operative dosing through to hospital discharge
To determine the safety of oral sildenafil to treat increased mPAP after cardiac surgery. | Begining 2 hours postoperatively through discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: David Mazer, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada